CLINICAL TRIAL: NCT03503903
Title: Efficacy of Wet Cupping on Reactive Oxygen Species and Antioxidant Capacity:A Self-controlled Interventional Study
Brief Title: Efficacy of Wet Cupping on Reactive Oxygen Species and Antioxidants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, SULEYMAN ERSOY, Asist.Prof. Department of Family Medicine, Karabuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBU-BAP-17/1-KA-070
Record Dates: First submitted 2018-04-04; First posted 2018-04-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: Wet cupping therapy; antioxidant capacity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wet Cupping (Experimental): One armed self-controlled study. Individuals in this arm will receive three concecutive WCT application
  Interventions: Procedure: Wet Cupping

INTERVENTIONS:
Procedure: Wet Cupping — CT was applied using plastic disposable vacuum cups on the back in the 5 areas of C7 cervical spine (DU14 acupoint), T2-4 lateral spine bilaterally (BL41-42 acupoint) and T6-8 lateral spine bilaterally (BL44-46), which are the recommended sites for headache (12). The cupping technique procedure was conducted in five phases:Primary suction,Area disinfection,Scarification,Secondary suction and bloodletting,Removing and dressing.

SUMMARY:
This study evaluates the efficacy of Wet cupping Therapy on oxidative stress and antioxidant capacity of the body.The healthy volunteers will receive wet cupping application and their initial venous blood samples and samples after the treatment will be evaluated for oxidative stress.

DETAILED DESCRIPTION:
Among the healthy individuals who applied for Wet Cupping Therapy (WCT) to Traditional and Complementary Therapies center in Karabuk Medical Faculty Education and Research Hospital for general wellbeing 24 volunteers were enrolled in the study. They will receive three concecutive WCT application in one month interval.Their venous blood samples obtained initially and after the completion of the three concecutive applications, will be evaluted in terms of Reactive Oxygen species and Antioxidant capacity.Additionally samples from the cupping blood during the first and the third WCT application will also be obtained and evaluated.

ELIGIBILITY:
Inclusion Criteria:

Healthy male adults

Must apply Traditional and complemantary medicine center for general well being.

Exclusion Criteria:

Any chronic disorder

Antiagregant drug usage

Bleeding disorders

-

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
TAS | 7 days
  Total antioxidant status
TOS | 7 days
  Total oxidant status

SECONDARY OUTCOMES:
SOD | 7 days
  Super oxide dismutase
CAT | 7 days
  Catalase

CONTACTS AND LOCATIONS:
Overall Officials: SULEYMAN ERSOY, Principal Investigator — Karabuk University
Locations (1):
- Karabuk University Karabuk Research and Education hospital, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] . Burton, M. Smith, T. Falkenberg, Building WHO's global strategy for traditional medicine, European Journal of Integrative Medicine 7(1) (2015) 13-15.
- [Background] M. Ahmedi, M.R. Siddiqui, The value of wet cupping as a therapy in modern medicine-An Islamic Perspective, (2014).
- [Background] S. El Sayed, H. Mahmoud, M. Nabo, Methods of wet cupping therapy (Al-Hijamah): in light of modern medicine and prophetic medicine, Alternative & Integrative Medicine (2013) 1-16.
- [Background] Sies H. Oxidative stress: oxidants and antioxidants. Exp Physiol. 1997 Mar;82(2):291-5. doi: 10.1113/expphysiol.1997.sp004024. PMID 9129943
- [Background] Lin MT, Beal MF. Mitochondrial dysfunction and oxidative stress in neurodegenerative diseases. Nature. 2006 Oct 19;443(7113):787-95. doi: 10.1038/nature05292. PMID 17051205
- [Derived] Ersoy S, Benli AR. Continue or stop applying wet cupping therapy (al-hijamah) in migraine headache:A randomized controlled trial. Complement Ther Clin Pract. 2020 Feb;38:101065. doi: 10.1016/j.ctcp.2019.101065. Epub 2019 Oct 18. PMID 31668556

DOCUMENTS (2):
  • Study Protocol (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT03503903/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT03503903/SAP_001.pdf